CLINICAL TRIAL: NCT06142630
Title: The Effects of Different Positions on the Diffusion and Blockade Effect of Ultrasound-guided Erector Spinae Plane Block
Brief Title: Different Positions on the Diffusion and Blockade Effect of Ultrasound-guided Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20230915-04
Record Dates: First submitted 2023-10-26; First posted 2023-11-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Erector Spinea Plane Block

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Supine group (No Intervention): Patients remained supine
- Prone group (Experimental): Patient remained prone
- Lateral position group (Experimental): Patient remained in a lateral position
  Interventions: Other: Alteration of patients' position after erector spinae plane block

INTERVENTIONS:
Other: Alteration of patients' position after erector spinae plane block — After the erector spinae plane block was completed, the patients kept supine, lateral or prone position according to the group allocated for 30 minute to ensure the spread of local anesthetic
  Arms: Lateral position group

SUMMARY:
After the completion of erector spinae plane block, the patient maintains different positions to assess the diffusion of local anesthetic and the effect of the block.

DETAILED DESCRIPTION:
Eighty-four patients were selected to undergo CT guided puncture localization of pulmonary nodules under local anesthesia, and the patients were divided into groups using a computer-generated random number in a ratio of 1:1:1. To ensure objectivity, a nurse who was not involved in the study prepared a sealed opaque envelope containing grouping information. Randomly divide patients into three groups: supine position group (S group, 28 patients), prone position group (P group, 28 patients), and lateral position group (L group, 28 patients). The patients underwent ultrasound guided ESPB on the puncture side before CT puncture localization. Ultrasound guided ESPB method: Using an ultrasound high-frequency linear array probe (5-13MHz, Sonosite, USA), the probe is placed parallel to the spine on the surface of the transverse process tip of the seventh thoracic vertebrae. Under ultrasound, the transverse process and spinal muscles are clearly exposed. Then, a short inclined plane puncture needle is used, and the needle is inserted from the head side using in-plane technology. After the needle tip reaches between the transverse process and erector spinae muscles, 1ml of physiological saline is injected using water separation technology to confirm the position of the needle tip, Then inject 30ml of local anesthetic solution (0.75% ropivacaine 15ml+iohexol 15ml). After the block was completed, patients in Group S remained in a supine position; Patients in group L maintained the blocking side above; Patients in Group P maintained a prone position. After 30 minutes of block completion, CT scan and puncture localization were performed, following with 3D reconstruction. The primary outcome was LA-contrast spread to the paravertebral space.The second outcomes were as follow: 1. spread to the neural foramina 2. cranio-caudal spread 3. spread to the epidural space 4. spread to the intercostal space.

ELIGIBILITY:
Inclusion Criteria:

Patients received CT guided puncture localization of pulmonary nodules under local anesthesia

Exclusion Criteria:

1. Allergic to local anesthetic
2. History of opioid abuse
3. Severe skin infection
4. Peripheral neuropathy
5. Dysfunction of blood coagulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence and number of local anesthetic diffusion segment into the paravertebral space | 30 minute after completion of the ESPB block
  Observation of local anesthetic spread spread into the paravertebral space with CT by a researcher who was blinded to group allocation

SECONDARY OUTCOMES:
Diffusion of local anesthetic into intercostal space | 30 minute after completion of the block
  The diffusion of local anesthetics to intercostal space was observed with CT by a researcher who was blinded to group allocation
Diffusion of local anesthetic into the epidural space | 30 minute after completion of the block
  Incidence and segment of local anesthetic spread into the epidural was assessed by a researcher who was blinded to group allocation
Sensory loss of cold | 30 minute immediately after completion of the nerve block
  The extent of sensory loss was assessed with cold stimulation, including the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall (paraspinal zone) by a researcher who was blinded to group allocation

CONTACTS AND LOCATIONS:
Overall Officials: Gu Jianping, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Munoz F, Cubillos J, Bonilla AJ, Chin KJ. Erector spinae plane block for postoperative analgesia in pediatric oncological thoracic surgery. Can J Anaesth. 2017 Aug;64(8):880-882. doi: 10.1007/s12630-017-0894-0. Epub 2017 Apr 26. No abstract available. PMID 28447318
- [Background] Ueshima H, Otake H. RETRACTED: Erector spinae plane block provides effective pain management during pneumothorax surgery. J Clin Anesth. 2017 Aug;40:74. doi: 10.1016/j.jclinane.2017.04.016. Epub 2017 Apr 28. No abstract available. PMID 28625453
- [Derived] Shan T, Zhang X, Zhao Z, Zhou X, Bao H, Su C, Tan Q, Han L, Yin J. Spread of local anaesthetic after erector spinae plane block: a randomised, three-dimensional reconstruction, imaging study. Br J Anaesth. 2025 Mar;134(3):830-838. doi: 10.1016/j.bja.2024.10.046. Epub 2025 Jan 8. PMID 39788818